CLINICAL TRIAL: NCT03789123
Title: Effects of Dienogest and Dienogest Plus Estradiol Valerate on Ovarian Reserve and Endometrioma Size
Brief Title: Effects of Dienogest and Dienogest Plus Estradiol Valerate in Ovarian Endometrioma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Collaborators: Kocaeli Derince Education and Research Hospital (Other); Suleymaniye Birth And Women's Health Education And Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.11.1.01.082.r1.101
Record Dates: First submitted 2018-11-22; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Ovarian Reserve
Keywords: Endometrioma; Estradiol valerate + dienogest; Dienogest; Ovarian reserve
MeSH Terms: conditions — Endometriosis | interventions — estradiol valerate-dienogest; dienogest

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (patients with OMA) (Experimental): I) Untreated patients (n=142)
  II) Dienogest (n=142)
  III) Dienogest/Estradiol valerate+Dienogest (n=142)
  Interventions: Drug: Estradiol valerate/dienogest
- Control Group(patients without OMA) (Sham Comparator): I) Untreated patients (n=142)
  II) Dienogest/Estradiol valerate+Dienogest (n=142)
  Interventions: Drug: Estradiol valerate/dienogest

INTERVENTIONS:
Drug: Estradiol valerate/dienogest — The effects of drugs given for endometrioma and contraception will be observed on ovarian reserve, endometrioma size and pain score.
  Other Names: Dienogest

SUMMARY:
Progesterone resistance in endometriosis is a known fact. The progestin derivatives used in endometriosis cause decidualization and atrophy of ectopic foci. Moreover, they inhibit neo-angiogenesis, provide suppress expansile/destructive growth facilitated by matrix metalloproteinases, and implantation of ectopic foci. The effect of drugs containing the estrogen-progesterone combination is mainly based on the inhibition of ovulation, decidualization and atrophy of ectopic foci. In estrogen-progesterone mechanism, it is known that estrogen has a progesterone receptor-enhancing effect, which may make progesterone more potent. Based on this, the investigators hypothesized that estrogen added to progesterone could lead to a further reduction in endometrioma size by various mechanisms which probably include the increased progesterone sensitivity in endometriosis. In addition, the investigators hypothesized that this therapy can alleviate the destructive effect of endometriomas on the ovarian reserve.

ELIGIBILITY:
Inclusion Criteria:

1. Study Group: At least one endometrioma greater than 3 cm, between 18-40 years of age, without surgical indication at the time of diagnosis, occasionally and intermittently controlled pain with NSAIDs or no pain symptom
2. Control Group: Patients with reproductive age without any ovarian cysts

Exclusion Criteria:

* suspicion of malignancy, irregular mentrual period, endocrine diseases, drug intake that may affect ovarian reserve in the last 6 months (i.e GnRH agonists), previous ovarian surgery, AMH levels under 2 ng/ml.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 710 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Ovarian reserve | up to 24 months
  The investigators evaluate serum anti-Müllerian hormone (AMH) level(ng/mL) using commercial elisa kits and antral follicle count (number) using ultrasonography. The patients with higher ovarian reserve represent a better outcome.

SECONDARY OUTCOMES:
Endometrioma Size | up to 24 months
  The investigators evaluate endometrioma size (centimeter) using ultrasonography.
Pain Score | up to 24 months
  Vas score (minimum score:0 and maximum score:10). The patients with lower pain scores represent a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Engin Oral, Prof.Dr. M.D, Study Director — Istanbul University Cerrahpasa Medical Faculty
Locations (1):
- Tolga Karacan, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided